CLINICAL TRIAL: NCT05709002
Title: A Fully Automated and Culturally-Adapted mHealth Intervention for Smoking Cessation Among Black Smokers With HIV
Brief Title: Smoking, Stress, HIV and Mobile Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Baylor College of Medicine (Other); University of Oklahoma (Other)
Responsible Party: Principal Investigator, Lorra Garey, Co-director of the RESTORE Lab, Research Assistant professor at the University of Houston, University of Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QKWEF8XLMTT3
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Cigarette Smoking
Keywords: HIV; Minority Stress; mHealth; Smoking Cessation; Anxiety Sensitivity
MeSH Terms: conditions — Cigarette Smoking; Smoking Cessation | interventions — Mannose-Binding Protein-Associated Serine Proteases; National Cancer Institute (U.S.)

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MASP+ app & NRT (Experimental): MASP+ is an intervention designed to assist Black smokers with HIV who experience elevated anxiety sensitivity to quit smoking through the use of educational videos, tailored messages, and interoceptive exercises designed to help the user overcome negative feelings of stress and nicotine withdrawal.
  Nicotine patches will be made available to provide adjunctive support.
  Interventions: Behavioral: MASP+
- QuitGuide app + NRT (Active Comparator): The QuitGuide app is a standard-of-care app that allows users to track nicotine cravings and provides motivational messages.
  Nicotine patches will be made available to provide adjunctive support.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: MASP+ — mHealth (mobile app) for smoking cessation
  Arms: MASP+ app & NRT
Behavioral: Control — A mobile app designed to assist the general population with smoking cessation.
  Other Names: National Cancer Institute (NCI) QuitGuide app
  Arms: QuitGuide app + NRT

SUMMARY:
The present investigation aims to address disparities in cigarette use outcomes among Black/African American adults with HIV. The specific aims of this study are: (1) To modify a recently developed, culturally adapted, mobile application for Black smokers by integrating information specifically relevant to Black persons with HIV/AIDS. (2) To conduct a randomized clinical trial for anxiety-sensitivity reduction and cigarette cessation among Black smokers with HIV.

DETAILED DESCRIPTION:
The current trial aims to refine and conduct a comprehensive cultural and HIV-sensitive adaptation of an initially tested, novel mobile intervention (MASP+) targeting anxiety sensitivity (AS) among Black/African American (daily) cigarette users with HIV/AIDS. The MASP+ app prompts users remotely throughout the day to assess mood symptoms, cigarette cravings or nicotine withdrawal symptoms, and general mental health. When respondents indicate they are struggling with cigarette urges or cravings, or if they are experiencing heightened levels of stress or anxiety, the app selects and delivers a tailored message from a library of messages and videos.

The MASP+ app has the potential to deliver highly effective and accessible treatment to a highly underserved subpopulation within the Black community considered to be at exceptionally high risk of smoking problems (social, psychological, physical) and smoking relapse.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infection (via self-report and picture of medication, lab tests, or diagnosis)
* 18+ years of age
* Self-identify as Black / African American
* Daily smoking (minimum of 10 cigarettes per day on average for at least 2 years)
* Motivated to quit smoking (≥ 5 on a 10-point scale)
* Willingness to discontinue cigarette use two weeks after baseline visit.
* English literacy (score of 4 or greater on REALM-SF)
* Moderate to high anxiety sensitivity (score of 5 or greater on SSASI)
* Provide a current picture of their cigarette package to verify smoking status
* Willing to complete all study surveys/assessments
* Agree to use nicotine replacement medications (NRT; nicotine patch and lozenges)
* Agree to attempt to quit smoking two weeks after completion of the baseline survey and receipt of study materials

Exclusion Criteria:

* Actively receiving (ongoing) pharmacotherapy or psychotherapy directly focused on the treatment of smoking cessation, and/or substance use, not provided by the study
* Non-fluent/limited English proficiency
* Self-reported pregnancy or intentions to become pregnant in near future
* Legal status that would interfere with participation
* Being non-Black
* Cognitive impairment (assessed via the 6-item Cognitive Impairment Test)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
Biochemically verified smoking abstinence | Weeks 1,2,3,4,5,6, & 28
  Our primary study outcome will be biochemically confirmed 7-day point prevalence abstinence 26 weeks following the scheduled quit day. The Bedfont iCO Smokerlyzer will be used to verify smoking status during the follow-up assessments. The monitors attach to the smartphone and will be used to remotely verify self-reported smoking abstinence during phone-based monitoring periods over the post-quit period. Our CO criteria for abstinence is consistent with numerous studies using cutoffs of < 7 ppm. This will be used to verify smoking status, as well as change in smoking behaviors throughout the study. As well, self-report measures of the Smoking History questionnaire (SHQ) will also be used to assess self-reported abstinence.

SECONDARY OUTCOMES:
Index of Engagement in HIV Care | Weeks 1 & 28
  The Index of Engagement in HIV Care is a brief (10-item) self-report measure of engagement in human immunodeficiency virus (HIV) care.
World Health Organization Quality of Life HIV (WHOQOL-HIV) | Weeks 1 & 28
  The WHOQOL-HIV questionnaire is composed of 36 items and is used to index quality of life among respondents living with HIV/AIDS.
ART Adherence | Weeks 1 & 28
  The Antiretroviral (ART) Adherence questionnaire is a brief scale used to assess frequency of missed ART medication doses and HIV care appointments among HIV+ patients/participants.

CONTACTS AND LOCATIONS:
Overall Officials: Lorra Garey, Ph.D., Principal Investigator — University of Houston; Michael Businelle, Ph.D., Principal Investigator — University of Oklahoma
Locations (1):
- Thomas Street at Quentin Mease Health Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bizier A, Jones A, Businelle M, Kezbers K, Hoeppner BB, Giordano TP, Thai JM, Charles J, Montgomery A, Gallagher MW, Cheney MK, Zvolensky M, Garey L. An Integrated mHealth App for Smoking Cessation in Black Smokers With HIV: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Apr 24;13:e52090. doi: 10.2196/52090. PMID 38657227